CLINICAL TRIAL: NCT06070519
Title: A Dynamic Evaluation of Chronic Heart Failure Prognosis: the MECKI Score
Acronym: MECKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Federico II University (Other); Fondazione Toscana Gabriele Monasterio (Other); The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CCM1827
Record Dates: First submitted 2023-10-02; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: HF - Heart Failure
Keywords: Cardiopulmonary exercise testing- CPET; Metabolic Exercise Cardiac Kidney Indexes (MECKI) score
MeSH Terms: conditions — Heart Failure | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sigle arm study (Experimental): HF patients who meets all the inclusion and none of the exclusion criteria
  Interventions: Diagnostic Test: CPET and related variables evaluation

INTERVENTIONS:
Diagnostic Test: CPET and related variables evaluation — At the baseline visit ,CPET-related variables, echocardiographic, ECG, therapy and blood chemistry data will be collected. The baseline CPET will be repeated within 2 weeks. Patients will perform 4 follow up visits at 6, 12, 18 and 24 months after the baseline visit. At every study step, it will be performed:
  * Echocardiography (LVEF)
  * Blood sample (Na+, MDRD, Hb)
  * Maximal ramp protocol CPET (peakVO2, VE/VCO2 slope)

SUMMARY:
The project is dedicated to the improvement of our capability to provide a precise and personalized prognosis in heart failure (HF) patients in stable conditions. The Metabolic Exercise test data combined with Cardiac and Kidney Indexes (MECKI) score is one of the 3 HF prognostic models recommended by the 2021 European HF guidelines and it is considered the most powerful prognostic tool available. MECKI score integrates cardiopulmonary exercise test (CPET) data with easy-to-obtain clinical, laboratory, and echocardiographic variables. It is based on 6 parameters: peak oxygen intake (peakVO2), minute ventilation/carbon dioxide production (VE/VCO2 slope), hemoglobin (Hb), Left Ventricle Ejection Fraction (LVEF), kidney function by Modification of Diet in Renal Disease (MDRD) formula, and sodium (Na+).

The aim of the present project is to assess the day-by-day MECKI score variability, CPET parameters interobserver variability, characterization of HF patients who change MECKI score values in 6 and 12 months, and the prognostic meaning of time dependent MECKI score changes.

DETAILED DESCRIPTION:
This is a low-intervention multicenter clinical trial aim at evaluating the role of time dependent prognostic parameters changes, moving from the single shot evaluation to dynamic analysis. Each participant center will perform patients' recruitment and follow up. At the baseline visit, CPET-related variables, echocardiographic, ECG, therapy and blood chemistry data will be collected. The baseline CPET will be repeated within 2 weeks. Patients will perform 4 follow up visits at 6, 12, 18 and 24 months after the baseline visit. At every study step, study procedures aimed to calculate MECKI score will be performed:

* Echocardiography (Left Ventricle Ejection Fraction - LVEF)
* Blood sample (Na+, MDRD, Hb)
* Maximal ramp protocol CPET (peakVO2, minute ventilation/carbon dioxide production (VE/VCO2) slope - VE/VCO2 slope)

ELIGIBILITY:
Inclusion Criteria:

* Previous or present HF symptoms (NYHA functional class I-IV, stage B and C of ACC/AHA classification)
* history or presence of left ventricular ejection fraction (LVEF)<40%
* unchanged HF medications for at least three months
* ability to perform a CPET
* no major cardiovascular treatment or intervention scheduled

Exclusion Criteria:

* History of pulmonary embolism
* moderate-to-severe aortic and mitral stenosis
* pericardial disease
* severe obstructive lung disease
* exercise-induced angina
* significant ECG alterations, or presence of any clinical comorbidity interfering with exercise performance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Day-by-day variability of MECKI score | through study completion, an average of 3 year
  Day by day variability of MECKI score will be done by comparing MECKI score value obtained at study run-in (day 0) and in a second evaluation of MECKI score performed within 2 weeks.
Identification of interobserver variability | through study completion, an average of 3 year
  CPET interobservers variability will be done by assessing CPET analysis done by two recognized CPET experts blinded on patients data

SECONDARY OUTCOMES:
Time-related dynamic changes of peak oxygen intake (VO2) | through study completion, an average of 3 year
  Modifications in peak oxygen intake (VO2) in 6-12-18-24 months will be evaluated in relation to prognosis
Time-related dynamic changes of minute ventilation/carbon dioxide production (VE/VCO2) slope | through study completion, an average of 3 year
  Modifications in minute ventilation/carbon dioxide production (VE/VCO2) slope in 6-12-18-24 months will be evaluated in relation to prognosis
Time-related dynamic changes of MDRD | through study completion, an average of 3 year
  Modifications of MDRD in 6-12-18-24 months will be evaluated in relation to prognosis
Time-related dynamic changes of LVEF | through study completion, an average of 3 year
  Modifications of LVEF in 6-12-18-24 months will be evaluated in relation to prognosis
Time-related dynamic changes of hemoglobin | through study completion, an average of 3 year
  Modifications of hemoglobin in 6-12-18-24 months will be evaluated in relation to prognosis
Time-related dynamic changes of Na+ | through study completion, an average of 3 year
  Modifications of Na+ in 6-12-18-24 months will be evaluated in relation to prognosis
The identification of the prognostic meaning of MECKI score changes at 6 months | 6 months
  Modifications of MECKI score at 6 months will be evaluated in relation to prognosis
The identification of the prognostic meaning of MECKI score changes at one year | one year
  Modifications of MECKI score at one year will be evaluated in relation to prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Piergiuseppe Agostoni, Prof, Principal Investigator — IRCCS Centro Cardiologico Monzino
Locations (4):
- Italy (4):
  - IRCCS Centro Cardiologico Monzino, Milan, Milan
  - Università di Napoli Federico II, Napoli
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Fondazione Toscana Gabriele Monasterio per la ricerca medica e di sanità pubblica, Pisa

REFERENCES:
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Agostoni P, Corra U, Cattadori G, Veglia F, La Gioia R, Scardovi AB, Emdin M, Metra M, Sinagra G, Limongelli G, Raimondo R, Re F, Guazzi M, Belardinelli R, Parati G, Magri D, Fiorentini C, Mezzani A, Salvioni E, Scrutinio D, Ricci R, Bettari L, Di Lenarda A, Pastormerlo LE, Pacileo G, Vaninetti R, Apostolo A, Iorio A, Paolillo S, Palermo P, Contini M, Confalonieri M, Giannuzzi P, Passantino A, Cas LD, Piepoli MF, Passino C; MECKI Score Research Group. Metabolic exercise test data combined with cardiac and kidney indexes, the MECKI score: a multiparametric approach to heart failure prognosis. Int J Cardiol. 2013 Sep 10;167(6):2710-8. doi: 10.1016/j.ijcard.2012.06.113. Epub 2012 Jul 15. PMID 22795401
- [Background] Agostoni P, Paolillo S, Mapelli M, Gentile P, Salvioni E, Veglia F, Bonomi A, Corra U, Lagioia R, Limongelli G, Sinagra G, Cattadori G, Scardovi AB, Metra M, Carubelli V, Scrutinio D, Raimondo R, Emdin M, Piepoli M, Magri D, Parati G, Caravita S, Re F, Cicoira M, Mina C, Correale M, Frigerio M, Bussotti M, Oliva F, Battaia E, Belardinelli R, Mezzani A, Pastormerlo L, Guazzi M, Badagliacca R, Di Lenarda A, Passino C, Sciomer S, Zambon E, Pacileo G, Ricci R, Apostolo A, Palermo P, Contini M, Clemenza F, Marchese G, Gargiulo P, Binno S, Lombardi C, Passantino A, Filardi PP. Multiparametric prognostic scores in chronic heart failure with reduced ejection fraction: a long-term comparison. Eur J Heart Fail. 2018 Apr;20(4):700-710. doi: 10.1002/ejhf.989. Epub 2017 Sep 26. PMID 28949086
- [Background] Paolillo S, Veglia F, Salvioni E, Corra U, Piepoli M, Lagioia R, Limongelli G, Sinagra G, Cattadori G, Scardovi AB, Metra M, Senni M, Bonomi A, Scrutinio D, Raimondo R, Emdin M, Magri D, Parati G, Re F, Cicoira M, Mina C, Correale M, Frigerio M, Bussotti M, Battaia E, Guazzi M, Badagliacca R, Di Lenarda A, Maggioni A, Passino C, Sciomer S, Pacileo G, Mapelli M, Vignati C, Clemenza F, Binno S, Lombardi C, Filardi PP, Agostoni P; MECKI Score Research Group (see Appendix). Heart failure prognosis over time: how the prognostic role of oxygen consumption and ventilatory efficiency during exercise has changed in the last 20 years. Eur J Heart Fail. 2019 Feb;21(2):208-217. doi: 10.1002/ejhf.1364. Epub 2019 Jan 11. PMID 30632680
- [Background] Salvioni E, Bonomi A, Re F, Mapelli M, Mattavelli I, Vitale G, Sarullo FM, Palermo P, Veglia F, Agostoni P. The MECKI score initiative: Development and state of the art. Eur J Prev Cardiol. 2020 Dec;27(2_suppl):5-11. doi: 10.1177/2047487320959010. PMID 33238744